CLINICAL TRIAL: NCT07053501
Title: The Effect of a Urinary Catheter Carrying Bag on Patients' Satisfaction, Body Image, Self-Esteem, and Shame: A Randomized Controlled Trial
Brief Title: Effect of a Urinary Catheter Carrying Bag on Satisfaction, Body Image, Self-Esteem, and Shame
Acronym: UCCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahar Ciftci (Other)
Responsible Party: Sponsor-Investigator, Bahar Ciftci, Assistant Professor, Department of Fundamental of Nursing, Atatürk University, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/513
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Long-Term Urinary Catheterization; Patient Satisfaction; Psychosocial Impact of Catheter Use; Low Self-Esteem; Body Image Disturbance
Keywords: Patient Satisfaction; Nursing Intervention; Self-Esteem Shame; Body Image; Catheter Carrying Bag; Urinary Catheter
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients used a specially designed urinary catheter carrying bag for 21 days along with training.
  Interventions: Device: Urinary Catheter Carrying Bag Use
- Control (No Intervention): Patients received routine catheter care without any intervention.

INTERVENTIONS:
Device: Urinary Catheter Carrying Bag Use — A wearable catheter carrying bag was provided to participants. It was designed to conceal the urine bag and increase comfort, privacy, and psychosocial well-being. Participants received training on its use and wore it during all daily activities for 21 days.
  Arms: Intervention

SUMMARY:
This study aimed to evaluate the impact of using an innovative urinary catheter carrying bag on the psychosocial well-being of patients who require long-term catheterization. The bag was designed to increase comfort, hygiene, and privacy by concealing the urine bag and minimizing potential embarrassment during daily activities.

A total of 70 patients who had been using an indwelling urinary catheter for at least three weeks were randomly assigned to either an intervention or a control group. The intervention group received a specially designed catheter carrying bag along with training on how to use it, while the control group received standard care without the carrying bag. All participants were monitored over a 21-day period.

Validated assessment tools were used to measure patient satisfaction, body image, self-esteem, and feelings of external shame at baseline and after the intervention period. The study was designed to explore whether the use of the catheter carrying bag could influence these psychosocial outcomes in individuals undergoing long-term catheterization.

This randomized controlled trial was conducted to inform future supportive care practices and explore non-pharmacological interventions that address both the physical and psychosocial needs of patients with indwelling urinary catheters.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted between July and December 2023 in the Emergency and Urology departments of X State Hospital. The aim was to investigate the effects of an innovative urinary catheter carrying bag (UCCB) on patients' psychosocial outcomes, including satisfaction, body image, self-esteem, and feelings of shame.

Participants (n=70) were adults aged 18 and older who had been using an indwelling urinary catheter for at least three weeks. Following ethical approval and informed consent, they were randomly assigned to intervention or control groups. The intervention group received a urinary catheter carrying bag along with detailed training, while the control group continued with standard care.

Data collection tools included the Patient Satisfaction-VAS, Body Image Scale, Rosenberg Self-Esteem Scale, and The Other as Shamer Scale. Assessments were conducted before the intervention and after the 21-day follow-up period.

Statistical analyses revealed that patients using the UCCB showed significantly greater improvements in all primary outcomes compared to the control group. Regression models confirmed that the carrying bag had a significant positive effect on patient satisfaction and self-esteem, and a significant negative effect on body image disturbance and shame.

This study provides empirical evidence that a simple, low-cost supportive device can positively influence the psychological well-being of catheter users. The findings suggest that integrating such tools into standard nursing protocols may improve holistic patient care.

ELIGIBILITY:
* Inclusion Criteria:
* Individuals aged 18 years or older
* Patients with an indwelling urinary catheter in place for at least 3 weeks
* Ability to communicate and provide informed consent
* Willingness to participate and comply with study procedures
* Exclusion Criteria:
* Patients with cognitive impairment or communication difficulties
* Presence of active urinary tract infection at the time of enrollment
* Severe physical or psychiatric condition interfering with participation
* Previous participation in a similar catheter-related intervention study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Satisfaction Score | Baseline and Day 21
  Patient satisfaction was assessed using a visual analog scale (VAS) at baseline (prior to intervention) and on Day 21 (post-intervention). The aim was to evaluate the impact of the catheter carrying bag on satisfaction related to urinary catheter use.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ State Hospital, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No